CLINICAL TRIAL: NCT00104754
Title: Phase II Trial of Liposome Encapsulated SN38 (LE-SN38) in the Treatment of Small Cell Lung Cancer
Brief Title: Liposomal SN-38 in Treating Patients With Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0322; CDR0000415847 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma

ARMS (1):
- liposomal SN-38 (Experimental): Patients receive SN-38 liposome IV over 90 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response or patients with stable disease (SD) who were previously treated before study enrollment receive up to 4 additional courses of treatment. Patients with CNS-only disease progression receive whole brain radiotherapy (WBRT). After completion of WBRT, these patients also receive up to 4 additional courses of treatment. Patients with disease progression to sites other than the CNS or patients with SD who were previously untreated before study enrollment are removed from the study.
  Quality of life is assessed at baseline, before each treatment course, and then annually for 3 years.
  After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 2 years.
  Interventions: Drug: liposomal SN-38

INTERVENTIONS:
Drug: liposomal SN-38

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal SN-38, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well liposomal SN-38 works in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with small cell lung cancer treated with SN-38 liposome that is dosed according to a UGT1A1-specific genotype.
* Determine the toxicity of this drug in these patients.
* Determine, preliminarily, overall and progression-free survival of patients treated with this drug.
* Determine the quality of life of patients treated with this drug.
* Correlate UGT1A1-specific haplotypes with toxicity of this drug in these patients.
* Correlate UGT1A1-specific haplotypes with outcomes of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to length of time since prior treatment (previously untreated disease OR chemosensitive disease and ≥ 3 months since prior treatment vs refractory disease OR chemoresistant disease and < 3 months since prior treatment).

Patients receive SN-38 liposome IV over 90 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response or patients with stable disease (SD) who were previously treated before study enrollment receive up to 4 additional courses of treatment. Patients with CNS-only disease progression receive whole brain radiotherapy (WBRT). After completion of WBRT, these patients also receive up to 4 additional courses of treatment. Patients with disease progression to sites other than the CNS or patients with SD who were previously untreated before study enrollment are removed from the study.

Quality of life is assessed at baseline, before each treatment course, and then annually for 3 years.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 73 patients (40 for stratum I and 33 for stratum II) will be accrued for this study within 16-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer meeting 1 of the following criteria:

  * Previously untreated disease

    * Extensive stage disease, as defined by any of the following:

      * Metastatic disease outside of the chest
      * Contralateral supraclavicular or contralateral hilar nodes that cannot be included in a single radiation port
      * Malignant pleural effusion
  * Previously treated disease

    * Limited or extensive stage disease
* Measurable disease

  * Lesions ≥ 1 cm and < 2 cm must be measured by spiral CT scan for pre- and post-treatment tumor assessment
* UGT1A1*28 genotype wt/wt (6/6 promoter TA repeats) OR wt/*28 (6/7 promoter TA repeats)

  * No *28/*28 (7/7 promoter TA repeats) genotype
* No mixed histology
* No uncontrolled CNS metastasis

  * Previously treated, stable CNS metastasis allowed
* No superior vena cava syndrome
* No malignant pericardial effusion
* No near obstruction of the trachea or main stem bronchi

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Total bilirubin < 1.5 times upper limit of normal (ULN) OR
* Direct bilirubin normal

Renal

* Creatinine < 1.5 times ULN

Cardiovascular

* No unstable angina pectoris
* No uncontrolled congestive heart failure
* No myocardial infarction within the past 3 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No syndrome of inappropriate antidiuretic hormone secretion
* No ectopic adrenocorticotrophic syndrome
* No Lambert-Eaton myasthenic syndrome
* No other severe paraneoplastic syndrome
* No active infection requiring oral or parenteral antibiotics
* No other life threatening disease
* No other malignancy except basal cell or squamous cell skin cancer, localized prostate cancer, superficial bladder cancer, or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF) during course 1 of study treatment

Chemotherapy

* No more than 1 prior chemotherapy regimen for this malignancy

  * Prior cyclophosphamide, doxorubicin, and vincristine (CAV) alternating with etoposide and cisplatin (EP) allowed
* More than 21 days since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 14 days since prior radiotherapy
* Concurrent palliative radiotherapy allowed except radiotherapy to a solitary measured index lesion

Surgery

* More than 21 days since prior major surgery

Other

* No other concurrent treatment for this malignancy
* No other concurrent investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Tumor response measured by number of responses | Up to 3 years

SECONDARY OUTCOMES:
Time to disease progression | Up to 3 years
Survival time | Up to 3 years
Change in quality of life (QOL) score over time | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James R. Jett, MD, Study Chair — Mayo Clinic